CLINICAL TRIAL: NCT00677703
Title: The Effect of Text Message Reminders on Contraceptive Continuation, a Randomized Controlled Trial
Brief Title: Txt Now 2 Decrease Pregnancies L8r: A Study to Evaluate the Effect of Daily Text Message Reminders on Pill Continuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Paula Castano, Assistant Clinical Professor, Columbia University
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: AAAC1600
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Contraceptives, Oral
Keywords: birth control pills; contraception; continuation; text messaging; contraceptive continuation; contraceptive knowledge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Participants will receive standard care without daily reminders.
- Text Messages (Experimental): Participants will receive a daily text message reminder for 6 months
  Interventions: Other: Daily Text Messages

INTERVENTIONS:
Other: Daily Text Messages — Text message reminders to take oral contraception daily:
  Each text message will be a short educational message listing the benefits of contraceptive use and providing instructions for avoiding common medication errors.
  Other Names: Text Messaging
  Arms: Text Messages

SUMMARY:
Teen girls and young women taking birth control pills may forget to take their pills or may stop taking them altogether. This places them at risk for unintended pregnancies. Most young women own cell phones and use them for text messaging. We will test whether contraceptive continuation is affected after six months of daily text message reminders.

DETAILED DESCRIPTION:
In 2000, there were 84 pregnancies for every 1,000 women aged 15 to 19 in the US (4). More than 90% of the resulting 900,000 teen pregnancies were unintended (6). Nationwide, teen pregnancy rates have dropped 28% since their peak in 1990 but dropped only 15% in Hispanic teens (4). New York state ranks 38th in the nation with 91 teen pregnancies per 1,000 teens. For Whites the teen pregnancy rate is only 52. Teen pregnancy rates are two to three times higher in Hispanics (130 pregnancies) and African Americans (167 pregnancies)(4). In New York City, the teen pregnancy rate is 99, even higher than the NY state and US rates (8).

Unintended pregnancy has long-term consequences that can disproportionately affect teens. Teen pregnancy negatively affects a teen's socioeconomic status. Pregnant teens are less likely to finish their education, more likely to be single parents and less likely to acquire work experience (9). Teen pregnancies are more likely to be medically complicated, with higher maternal and infant morbidity and mortality rates than in older pregnant women (10). Over one third of teen pregnancies end in abortion. Once a teen has one delivery, she is at increased risk to have another. Furthermore, a daughter of a teen pregnancy is more likely to have a teen pregnancy herself (11). Consistent contraceptive use is the only way to prevent pregnancy (and all of its consequences) in sexually-active teens. In a study of OC use in our population, 99% of the pregnancies that did occur were in women who had discontinued their OC during the study period (1).

The National Survey of Family Growth, a nationwide study examining contraceptive use in 2,271 teenagers, showed that 98% of sexually-active teenagers had used a contraceptive method at some time (12). Among teen contraceptors, 53% use oral contraceptives (OC) - the highest percentage among all age groups (12). The percentage of African American and Hispanic teens using contraception is lower than white teens (12). The World Health Organization estimates that half of patients take their medication improperly (13). One million of the United States' unintended pregnancies result from improper OC use, failure or discontinuation (14). Teens discontinue OCs because they experience side effects, misunderstand instructions for use and do not establish a pill-taking routine (3). In a study of OC use in inner city family planning clinics, we found discontinuation rates of 40% and 61% at three and six months, respectively (1). For the 595 teens in that study, discontinuation rates were 53% and 75% at three and six months, respectively. High discontinuation rates are also reported elsewhere (15-19). Improving OC continuation in the U.S. by just 10% can lead to a 7% reduction in unintended pregnancies and an annual savings of $280 million (1995 dollars) (14). Nationally, that could mean a reduction of unintended teen pregnancies by 63,000.

Wireless text messaging is a technology that was effective in improving medication adherence in clinical trials of vaccines and smoking cessation in Spain and South Africa (20,21). Text messaging has also been found to be more effective than telephone call-backs and scheduled clinic revisits in providing patients in London with lab results and decreasing the time for them to return to clinic for treatment (22). Cell phones have more recently become widespread in America and cell phone use continues to increase. A 2005 survey of wireless providers revealed that there were nearly 208 million wireless subscribers in the US, nearly 26 million more than in 2004 (23). Americans use cell phones for more than talking; they can use the text message function to share photos, to vote for reality television programming contestants, to receive daily jokes or to receive ring tones. Sixty-four percent of teens with cell phones use text messaging (24). Urban teen girls are more likely to use text messaging than boys or adults (24).

To assess cell phone use in our own population we carried out a survey of 2,521 racially-diverse reproductive-aged women, including 473 teens, attending family planning clinics in NYC. Cell phone usage was 77% among teens, and 81% of them read and send text messages (5). One-third of the participants in this feasibility survey worry about forgetting to take their medications and 30% would like to receive text message reminders for this (5). There are no studies of the effectiveness of text message reminders on contraceptive continuation rates.

Successful teen pregnancy prevention programs use varied, multifactorial approaches (2). We propose a study using an existing technology, text messaging, in an innovative way to improve OC continuation rates. Daily text messages will provide information regarding side effects, their management and instructions for troubleshooting common pill-taking mistakes. They may also help teens and young women establish a dosing routine.

ELIGIBILITY:
Inclusion Criteria:

* aged <25 years requesting OC as their primary method of contraception
* currently sexually active or anticipating sexual activity within the next 30 days
* owns cell phone with text messaging capability

Exclusion Criteria:

* contraindications to combined hormonal contraception per clinic protocol (e.g., hypertension)
* previous participation in this study

Max Age: 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 968 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
contraceptive continuation | 6 months

SECONDARY OUTCOMES:
change in contraceptive knowledge scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Castano, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Planned Parenthood Boro Hall, Brooklyn, New York, United States

REFERENCES:
- [Background] Castano PM, Martinez RA. Harnessing technology for adolescent health promotion. Adolesc Med State Art Rev. 2007 Aug;18(2):400-6, xiii. PMID 18605654
- [Result] Castano PM, Westhoff C, Andres Martinez R, Lara M. The effect of daily text message reminders on adolescent oral contraceptive pill continuation. Journal of Adolescent Health 44(2): S17, 2009.
- [Result] Hall KS, Westhoff CL, Castano PM. The impact of an educational text message intervention on young urban women's knowledge of oral contraception. Contraception. 2013 Apr;87(4):449-54. doi: 10.1016/j.contraception.2012.09.004. Epub 2012 Oct 10. PMID 23062523
- [Result] Castano PM, Bynum JY, Andres R, Lara M, Westhoff C. Effect of daily text messages on oral contraceptive continuation: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):14-20. doi: 10.1097/AOG.0b013e31823d4167. PMID 22143257